CLINICAL TRIAL: NCT00482794
Title: Genetics of Antiphospholipid Antibody Syndrome
Brief Title: Genetic Risk Factors Associated With Antiphospholipid Antibody Syndrome
Acronym: APS
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00013845
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid Antibody Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, and DNA samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Individuals with APS who also have one or more of their family members affected specifically by APS
- 2: Individuals with APS who also have one or more of their family members affected by another type of autoimmune disorder, such as lupus or rheumatoid arthritis.
- 3: Individuals with APS and no family or no family affected with APS or another autoimmune disorder

SUMMARY:
Antiphospholipid antibody syndrome (APS) is characterized by the presence of antiphospholipid antibodies, which are proteins in the blood that interfere with the body's ability to perform normal blood clotting. Clinical problems associated with antiphospholipid antibodies include an increased risk for the formation of blood clots in the lungs or deep veins of the legs, stroke, heart attack, and recurrent miscarriages. It is possible that some people with APS have a genetic predisposition for developing the syndrome. This study will use a genetic strategy to identify potential inherited risk factors for the development of APS by recruiting people with APS who have family members also affected by the syndrome or by another autoimmune disorder, such as lupus or rheumatoid arthritis.

DETAILED DESCRIPTION:
APS is an autoimmune disorder that causes an increased risk for developing a venous or arterial thromboembolism, as well as recurrent miscarriages. APS frequently occurs in people with lupus, and is referred to as secondary APS in this case. Many people who have APS, however, do not have another autoimmune disorder, and their disease is referred to as primary APS. APS may be a genetic disorder, and identifying the gene(s) that predisposes an individual to develop it could lead to a better understanding of the disease, as well as improved therapies. This study will use a genetic strategy to identify potential risk factors for the development of APS by recruiting people with APS who have family members who are either affected by the syndrome or who have another autoimmune disorder. The results of the genetic testing will be compared among the following two groups of families: people with APS who also have one or more of their family members affected specifically by APS; and people with APS who also have one or more of their family members affected by another type of autoimmune disorder, such as lupus or rheumatoid arthritis.

Participants in this study will perform a pre-screening questionnaire over the phone to determine relevant clinical diagnoses and collect a brief family history of autoimmune disorders. Eligible participants will receive an enrollment package in the mail. If possible, participants will then report to the study site to supply a detailed family and medical history and provide a blood sample for analysis for antiphospholipid antibodies and preparation of genomic DNA. If participants are unable to attend the study visit, the interviews will be conducted over the phone. Those who are unable to attend the site visit will receive a blood enrollment kit in the mail, and these participants will report to a convenient location for phlebotomy services. Participants who have already provided blood samples for the APS Collaborative Registry (APSCORE) may not have to provide another sample for this study. Information collected for statistical analysis will include the following data: demographic information; co-morbid conditions and chronic risk factors; lipid profile; history of recurrent infections, renal failure, and cardiovascular disease; height and weight; details of any medications and supplements currently being taken; venous and arterial thromboembolic events; and any history of adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Persistent presence of an antiphospholipid antibody, as defined by one or both of the following criteria:

  1. Medium or high anticardiolipin antibody level in the blood on two or more occasions at least 6 weeks apart
  2. Presence of lupus anticoagulant in the plasma on two or more occasions at least 6 weeks apart
* Presence of clinical symptoms seen in patients with APS, including vascular thrombosis (one or more clinical episodes of arterial, venous, or small vessel thrombosis in any tissue or organ) and/or pregnancy morbidity, defined as any of the following:

  1. One or more unexplained deaths of a morphologically normal fetus at or beyond the 10th week of gestation, with normal fetus morphology documented by ultrasound or direct examination or the fetus
  2. One or more premature births of a morphologically normal baby at or before the 34th week of gestation because of severe pre-eclampsia, eclampsia, or severe placental insufficiency
  3. Three or more unexplained consecutive spontaneous abortions before the 10th week of gestation, with maternal anatomic or hormonal abnormalities and paternal and maternal chromosomal causes excluded
* People who have elevated antiphospholipid antibody levels but do not fully meet clinical criteria for APS, and do have affected family members, will be considered for enrollment

Exclusion Criteria:

* No documented presence of antiphospholipid antibody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with antiphospholipid antibody syndrome and their family members
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2006-06; Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
characterize genetic risk factors associated with the development of familial antiphospholipid antibody syndrome. | duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Ortel, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine JS, Branch DW, Rauch J. The antiphospholipid syndrome. N Engl J Med. 2002 Mar 7;346(10):752-63. doi: 10.1056/NEJMra002974. No abstract available. PMID 11882732
- [Background] Cervera R, Piette JC, Font J, Khamashta MA, Shoenfeld Y, Camps MT, Jacobsen S, Lakos G, Tincani A, Kontopoulou-Griva I, Galeazzi M, Meroni PL, Derksen RH, de Groot PG, Gromnica-Ihle E, Baleva M, Mosca M, Bombardieri S, Houssiau F, Gris JC, Quere I, Hachulla E, Vasconcelos C, Roch B, Fernandez-Nebro A, Boffa MC, Hughes GR, Ingelmo M; Euro-Phospholipid Project Group. Antiphospholipid syndrome: clinical and immunologic manifestations and patterns of disease expression in a cohort of 1,000 patients. Arthritis Rheum. 2002 Apr;46(4):1019-27. doi: 10.1002/art.10187. PMID 11953980
- [Background] Scofield RH, Bruner GR, Kelly JA, Kilpatrick J, Bacino D, Nath SK, Harley JB. Thrombocytopenia identifies a severe familial phenotype of systemic lupus erythematosus and reveals genetic linkages at 1q22 and 11p13. Blood. 2003 Feb 1;101(3):992-7. doi: 10.1182/blood-2002-04-1003. Epub 2002 Sep 12. PMID 12393658
- [Background] Kelly JA, Thompson K, Kilpatrick J, Lam T, Nath SK, Gray-McGuire C, Reid J, Namjou B, Aston CE, Bruner GR, Scofield RH, Harley JB. Evidence for a susceptibility gene (SLEH1) on chromosome 11q14 for systemic lupus erythematosus (SLE) families with hemolytic anemia. Proc Natl Acad Sci U S A. 2002 Sep 3;99(18):11766-71. doi: 10.1073/pnas.182162399. Epub 2002 Aug 21. PMID 12192084
- [Background] Ortel TL. The antiphospholipid syndrome: what are we really measuring? How do we measure it? And how do we treat it? J Thromb Thrombolysis. 2006 Feb;21(1):79-83. doi: 10.1007/s11239-006-5581-x. PMID 16475047